CLINICAL TRIAL: NCT00626678
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Adjuvant Azathioprine Therapy in New Cases of Pemphigus Vulgaris Receiving Prednisone
Brief Title: Azathioprine Versus Placebo in Pemphigus Vulgaris Treated With Prednisolone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Cheyda Chams-Davatchi, Department of Dermatology, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 87- 01-30 - 6907
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus Vulgaris; Azathioprine; Prednisone
MeSH Terms: conditions — Pemphigus | interventions — Azathioprine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral administration of prednisone and azathioprine throughout study
  Interventions: Drug: Azathioprine; Drug: Prednisone
- 2 (Placebo Comparator): Oral administration of prednisone and placebo throughout study
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Azathioprine — It is given in a consistent dosage of 2.5 mg/kg/day throughout the study
  Other Names: Imuran
  Arms: 1
Drug: Prednisone — Oral corticosteroid initiated at 2 mg/kg/day dosage. Dosage may be tapered primarily by 1/3 total dosage if no new blister, then 5 mg every three days to reach the daily dosage of 30 mg then tapered by 1.25 mg every week to reach daily dosage of 20 mg/day, then tapered by 1.25 mg every two weeks to reach daily dosage of 10 mg, then tapered by 1.25 mg monthly to reach daily dosage of 7.5 mg and continue this dosage for six months then tapered to 5 mg/day if no new lesions are observed as determined by clinical assessment of the investigator.
  Other Names: Meticorten ®; Deltasone®; Orasone®
Drug: Placebo — Placebo given in place of Azathioprine 2.5 mg/kg/day throughout the study
  Other Names: Vehicle
  Arms: 2

SUMMARY:
Description: Pemphigus vulgaris is an autoimmune, chronic and recurrent blistering disease with unknown etiology that affects mucosa and skin of patients with significant morbidity and mortality.

The treatment back-bone is based on prednisolone administration. There are controversies on the opportunity of adding immunosuppressive drugs. For some, they are just corticosteroid sparing drugs. For others, they are disease modifying drugs.

The purpose of this trial is to compare efficacy and safety of azathioprine vs. placebo in new cases of pemphigus vulgaris treated with prednisolone.

DETAILED DESCRIPTION:
The purpose of this trial is to compare efficacy and safety of azathioprine vs. placebo in new cases of pemphigus vulgaris treated with prednisolone.

Official Title: Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Azathioprine in New Cases of Pemphigus Vulgaris Receiving Prednisolone

Randomized Double Blind Controlled Trial of Azathioprine versus Placebo in new cases of Pemphigus Vulgaris treated with Prednisolone

Study Type: Interventional

Study Design: Treatment, Randomized, Double Blind (Subject, Caregiver), Placebo Controlled, Parallel Assignment, Safety/Efficacy Study

Condition Intervention Phase Pemphigus Vulgaris Drug: Azathioprine Drug: Prednisolone Other: Placebo Phase II

ELIGIBILITY:
Inclusion Criteria:

* Lesions clinically consistent with pemphigus vulgaris
* Diagnosis confirmed by histology in terms of acantholysis within past month
* Positive DIF

Exclusion Criteria:

* Any nursing or pregnant woman
* Any history of chronic diseases including liver disease, Chronic Renal Failure, Chronic Heart Failure or Ischemic Heart Disease
* Present diagnosis of hepatitis confirmed by serology or elevated hepatic enzymes;
* Clinically significant concurrent medical disease or laboratory abnormalities evidenced by one or more of the following:
* Hepatobiliary AST or ALT ≥ 1.5 × upper limit of normal (ULN);alkaline phosphatase ≥ 1.5 × ULN; or, total bilirubin > 90% of the ULN;
* Renal serum creatinine > 1.5 mg/dL; or, significant proteinuria > 2+ on urinary dip test;
* Hematologic hemoglobin < 11 mg/dL; leukocytes < 3.5 × 109/L; neutrophils < 1.5 × 109/L; or, platelets < 100 × 109/L; Presence of anemia, leukopenia or thrombocytopenia
* Any sign of patient's non-compliance
* Known hypersensitivity to study drugs, prednisone or azathioprine
* Participating in another clinical trial at the time of screening and enrollment

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
• Disease activity index | Throughout study; first two weeks every day, then weekly for two weeks, then monthly for eleven months

SECONDARY OUTCOMES:
Total dose of corticosteroid | At the end of study
Occurence of any adverse event | Throughout study
Occurence of Grade 3 or higher treatment-related adverse event | Throughout study
Adverse events resulting in discontinuation and assessed by the investigators as at least possibly related to treatment | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Cheyda Chams-Davatchi, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Department of Dermatology, Tehran University of Medical Sciences, Tehran, Tehran Province, Iran